CLINICAL TRIAL: NCT03373253
Title: Treatment-Resistant Depression Cohort in Europe
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108384; 54135419DEP4001 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2017-12-08; First posted 2017-12-14 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Participants With Diagnosis of Depression: This study will evaluate participant's socio-demographic, disease-related and treatment-related characteristics along with outcomes in routine clinical practice across the European region. Only data available within clinical practice, through routine therapeutic procedures and diagnostic assessments, will be recorded. Individual participant information will be recorded from participant's medical records or by use of specific questionnaires.

SUMMARY:
The purpose of this study is to assess the participants socio-demographics and disease-related characteristics, long-term naturalistic treatment patterns and the clinical, social and economic outcomes of routine clinical practice in the treatment of participants with treatment-resistant depression (TRD) in a variety of European countries.

DETAILED DESCRIPTION:
This TRD cohort study will collect critically important data from routine clinical practice in Europe which will further substantiate the understanding of TRD in European clinical practice, with the aim of improving guidance and informing the development of better treatment strategies for this medically important condition. All data recorded in the case report form (CRF) should be documented in participants' medical records, that will be the primary data source of each participant. Participants who meet the diagnostic criteria for Major Depressive Disorder (MDD) and the diagnostic criteria for TRD, and are initiating or planned to initiate a new antidepressive treatment regimen will participate in the study. The end of the entire study will be 6 months after enrollment of the last participant in the study.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for single episode or recurrent MDD, without psychotic features, according to either the International Statistical Classification of Diseases and Related Health Problems, Tenth Revision (ICD-10) or the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Is considered to suffer from a moderate or severe depressive syndrome, as defined by a Montgomery-Asberg Depression Rating Scale (MADRS) total score greater than or equal to (>=) 20 at baseline
* Meets/has met the TRD criteria, defined as lack of clinically meaningful improvement, as indicated by a Clinical Global Impression-Change (CGI-C) score >= 4 and/or less than or equal to (<=) 25 percent (%) improvement in MADRS total score (lack of tolerability is not an indicator of non-response), with at least 2 different oral antidepressant treatments (of the same class, of a different class, or a combination of antidepressants or antidepressant with adjunctive antipsychotics) in the current episode of depression, prescribed in adequate dosages (as defined in the Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire [MGH ATRQ]) for adequate duration (at least 6 weeks) with adequate treatment adherence assessed by physicians
* Is initiating a new antidepressive treatment to treat the current depressive episode
* Must be capable of providing informed consent, based on the opinion of the participating physician

Exclusion Criteria:

* Has a current or prior diagnosis of a psychotic disorder, MDD with psychotic features, bipolar or related disorders, or intellectual disability, according to DSM-5 or ICD-10
* Has homicidal ideation/intent or has suicidal ideation with some intent to act, within 1 month prior to enrollment (per the physician's clinical judgment or based on the Columbia-Suicide Severity Rating Scale [C-SSRS] corresponding to a response of "Yes" on Item 4 [active suicidal ideation with some intent to act, without specific plan] or Item 5 [active suicidal ideation with specific plan and intent]) or a history of suicidal behavior within 1 year prior to enrollment
* Has a history of moderate or severe substance use disorder or severe alcohol use disorder according to DSM 5 criteria, except for nicotine and caffeine, within 6 months prior to enrollment
* Has a lifetime history of hallucinogen-related substance use disorder, with ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3,4 methylenedioxy-methamphetamine (MDMA)
* Has participated in or is currently enrolled in any clinical trial or observational study within the current episode
* Has previously received esketamine at any time

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Major Depressive Disorder (MDD) who fulfill the most commonly adopted criteria for treatment-resistant depression (TRD) with outcomes in routine clinical practice across the European region will be part of the study.
Sampling Method: Probability Sample
Enrollment: 830 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Resistant Depression (TRD) Participants With Change From Baseline in Socio-demographic Characteristics | Baseline up to 21 months (end of study)
  Number of TRD participants with change from baseline in socio-demographic characteristics (education, occupational status, living status, economic status, marital status, legal status) will be assessed.
Treatment Patterns Over Time for TRD Participants | Baseline up to 21 months (end of study)
  Treatment patterns (pharmacological and/or non-pharmacological) of TRD participants will be assessed over time.
Percentage of Participants With Disease-Related Characteristics | Up to 21 months
  Percentage of participants with disease-related characteristics for TRD among Major Depressive Disorder (MDD) participants will be assessed.
Severity of Symptoms as Measured by Montgomery-Asberg Depression Rating Scale (MADRS) | Up to 21 months
  The MADRS is a clinician-rated scale designed to measure changes in depression severity due to antidepressant treatment.The MADRS consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms) for a total possible score of 60. Higher scores represent a more severe condition.
Participant's Clinical Global Impression-Severity (CGI-S) Score | Up to 21 months
  The CGI-S evaluates the severity of psychopathology on a scale of 0 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants. The CGI-S permits a global evaluation of the participant's condition at a given time.
Participant's Clinical Global Impression-Change Scale (CGI-C) | Up to 21 months
  The CGI-C is a clinician-rated 7 point scale, ranging from 1 (very much improved) to 7 (very much worse). The CGI C scale will be used in this study to assess any improvement or worsening in a participant's condition versus previous assessments.
Healthcare Resource Utilization in TRD Participants | Up to 21 months
  Healthcare resources utilized in TRD participants will be estimated.
European Quality of Life (EuroQol) 5-Dimension 5-Level Questionnaire | Up to 21 months
  The EQ-5D-5L descriptive system comprises 5 dimensions - mobility, self-care, usual activities, pain/discomfort, and anxiety/depression - each of which is divided into 5 levels of perceived problems (Level 1 indicating no problem, Level 2 indicating slight problems, Level 3 indicating moderate problems, Level 4 indicating severe problems, and Level 5 indicating extreme problems).
Quality of Life in Depression Scale (QLDS) | Up to 21 months
  The QLDS is a disease-specific PRO used to document the impact that depression has on a participant's quality of life. The QLDS is a 34-item self-rated questionnaire consisting of dichotomous response questions, with responses being either True/Not True or Yes/No. It is scored binomially (that is, 0 or 1), with high scores on the QLDS indicating a lower quality of life.
Work Productivity and Activity Impairment (WPAI) | Up to 21 months
  The WPAI produces 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment. The WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Level of Disability as Sheehan Disability Scale (SDS) | Up to 21 months
  Participant-reported outcome of functional impact and associated disability will be documented by use of the SDS, a 5-item questionnaire. The first 3 items of the SDS document disruption of work/school, social life, and family life/home responsibilities, each using a rating from 0 to 10. The scores for the first 3 items are summed to create a total score of between 0 and 30, a higher score indicative of greater impairment. It also has 1 item on days lost from school or work and 1 item on days when underproductive.
Sequence of Treatments in Participants with TRD | Up to 21 months
  Treatment sequences for participants with TRD within routine clinical care in Europe will be assessed.
Demographic Characteristics of TRD Participants | Baseline
  Demographic characteristics (such as age and gender) of TRD participants will be assessed at baseline.
Suicidality Risk (Ideation and Attempts) as Measured by Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Baseline
  Suicidal ideation or behavior will be measured using C-SSRS score. C-SSRS is a clinician rated assessment of suicidal behavior and/ or intent. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 yes/no items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (98):
- Belgium (9):
  - Hauwaert An, Bilzen
  - AZ Sint-Lucas, Bruges
  - C.H.U. Brugmann, Brussels
  - Psy Pluriel-Pastur, Brussels
  - Psychiatrisch Centrum Dr Guislain, Ghent
  - CHU Sart Tilman, Liège
  - Hôpital du Petit Bourgogne, Liège
  - Clinique Saint Pierre, Ottignies
  - St-Andries Ziekenhuis, Tielt
- Germany (23):
  - Klinik f. Psychiatrie, Psychosomatik u Psychoth, Bamberg
  - Fliedner Klinik Berlin, Berlin
  - Praxis Dr. med. Jana Thomsen, Berlin
  - Charite Campus Benjamin Franklin, Berlin
  - Alexander Schulze - Germany, Berlin
  - Praxis Dr. med. Kirsten Hahn, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitatsklinikum Carl Gustav Carcus Dresden, Dresden
  - Kliniken Essen-Mitte, Essen
  - Klinikum der Johann Wolfgang Goethe -Universitaet, Frankfurt
  - Gemeinschaftspraxis F. Neurologie, Psychiatrie Und Psychotherapie Dres. Leonhardt U. Sallach, Gelsenkirchen
  - Asklepios Klinik Nord - Ochsenzoll, Hamburg
  - Privat-Nervenklinik, Dr. med. Kurt Fontheim - Germany, Liebenburg
  - Universitaetsklinikum Magdeburg A.oe.R, Magdeburg
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
  - Medizinisches Versorgungszentrum Mittweida - Germany, Mittweida
  - NPZR - Neuropsychatrisches Zentrum Riem, München
  - Johanniter Krankenhaus Oberhausen, Oberhausen
  - Praxis Kuehn, Oranienburg
  - Danuvius Klinik GmbH Pfaffenhofen, Pfaffenhofen
  - Somni Bene GmbH, Schwerin
  - Zentrum f. Neurologisch- Psychiatrische Studien und Begutachtung, Siegen
  - Praxis Dipl.-med. Stefan Kusserow, Stralsund
- Italy (22):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia Presidio Spedali Civili, Brescia
  - Azienda Ospedaliero Univ. Policlinico Gaspare Rodolico, Catania
  - Policlinico Universitario Germaneto, Catanzaro
  - Azienda Sanitaria 3 Genovese, Genova
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Casa di Cura Villa Von Siebenthal, Genzano di Roma
  - AUSL LE di Lecce, Lecce
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - Azienda Socio Sanitaria Territoriale di Monza Presidio San Gerardo, Monza
  - Azienda Ospedaliera Universitaria Maggiore della Carità, Novara
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda ospedaliera Sant'Andrea di Roma- Università di Roma La Sapienza, Roma
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Rome
  - Dipartimento Interaziendale di Salute Mentale, Siena
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette Di Ancona
- Netherlands (3):
  - Praktijk voor Psychiatrie en Psychotherapie, Heerde
  - Psychiatriepraktijk Helmind, Helmond
  - MAPTA Psychiatrie, Zeist
- Portugal (10):
  - Centro Hospitalar do Baixo Vouga E P E Unidade de Aveiro, Aveiro
  - Unidade Local de Saúde do Baixo Alentejo, EPE, Beja
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Hospital do Espirito Santo, EPE, Evora
  - Centro Hospitalar do Tâmega e Sousa, EPE - Hospital Padre Americo, Vale do Sousa, Guilhufe - Penafiel
  - Centro Hospitalar de Leiria, Leiria
  - Hospital CUF Inf. Santo, Lisbon
  - Fund. Champalimaud, Lisbon
  - Uls Santo Antonio - Hosp. Magalhaes Lemos, Porto
- Spain (16):
  - Hosp. Del Mar, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. de Bellvitge, Barcelona
  - Consulta Dr Salvador Sarro, Barcelona
  - Hosp. Gral. de Ciudad Real, Ciudad Real
  - Centro de Salud Mental Toscar, Elche
  - Hosp. Univ. de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Csm Fuencarral, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Puerta Del Sur, Móstoles
  - Centro Salud Mental La Corredoria, Oviedo
  - Hospital Psiquiátrico Provincial Rebullón, Pontevedra
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. de Torrevieja, Torrevieja
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. de Zafra, Zafra
- United Kingdom (15):
  - Royal Cornhill Hospital, Aberdeen
  - University of Bristol, Bristol
  - Surrey and Borders Partnership NHS Foundation Trust, Chertsey
  - West Park Hospital, Darlington
  - Royal Derby Hospital, Derby
  - Royal Edinburgh Hospital, Edinburgh
  - Burntwood and Lichfield CMHT, Lichfield
  - Institute of Psychiatry, London
  - Barnes-jewish Hospital, London
  - Berrywood Hospital, Northampton
  - Kingfisher Court, Radlett
  - Royal South Hants Hospital, Southampton
  - Cornwall Learning Disabilities Service, Truro
  - Westhaven Hospital, Weymouth
  - Vale House, Winsford

REFERENCES:
- [Derived] Oliveira-Maia AJ, Rive B, Godinov Y, Mulhern-Haughey S. Estimating the benefit of esketamine nasal spray versus real-world treatment on patient-reported functional remission: results from the ICEBERG study. Front Psychiatry. 2024 Oct 7;15:1459633. doi: 10.3389/fpsyt.2024.1459633. eCollection 2024. PMID 39435126
- [Derived] Oliveira-Maia AJ, Morrens J, Rive B, Godinov Y, Cabrieto J, Perualila N, Barbreau S, Mulhern-Haughey S. ICEBERG study: an indirect adjusted comparison estimating the long-term benefit of esketamine nasal spray when compared with routine treatment of treatment resistant depression in general psychiatry. Front Psychiatry. 2023 Oct 31;14:1250980. doi: 10.3389/fpsyt.2023.1250980. eCollection 2023. PMID 38025433
- [Derived] Oliveira-Maia AJ, Rive B, Morrens J, Godinov Y, Cabrieto J, Perualila N, Mulhern-Haughey S. Indirect adjusted comparison of 6-month clinical outcomes between esketamine nasal spray and other real-world polypharmacy treatment strategies for treatment resistant depression: results from the ICEBERG study. Front Psychiatry. 2023 Oct 31;14:1250987. doi: 10.3389/fpsyt.2023.1250987. eCollection 2023. PMID 38025416
- [Derived] Perugi G, Calo P, De Filippis S, Rosso G, Vita A, Adami M, Ascione G, Morrens J, Delmonte D. Clinical Features and Outcomes of 124 Italian Patients With Treatment Resistant Depression: A Real-World, Prospective Study. Front Psychiatry. 2021 Nov 5;12:769693. doi: 10.3389/fpsyt.2021.769693. eCollection 2021. PMID 34803777